CLINICAL TRIAL: NCT06909422
Title: A Mobile Intervention to Enhance Your Mood: A Test of the Acceptability and Efficacy
Brief Title: Mobile Thinking Intervention: A Inital Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lauren Luther, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013893; Internal Award (Other Grant/Funding Number: University of Alabama at Birmingham)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Clinical High Risk for Psychosis (CHR)
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Intervention to Target Biased Thinking (Experimental)
  Interventions: Behavioral: Mobile Intervention for Biased Thinking

INTERVENTIONS:
Behavioral: Mobile Intervention for Biased Thinking — This intervention will be delivered via a mobile application.

SUMMARY:
This study will test the inital efficacy of a brief mobile intervention targeting biased thinking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or related psychotic disorder OR
* Identified as being at clinical high risk for psychosis in symptom interviews

Exclusion Criteria:

* Recent changes in mental health treatment in past month or two months if on depot

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Defeatist Beliefs Scale - 15 | Measured at Baseline and post intervention (6 weeks)
  Measure of Defeatist Performance Beliefs
Brief Negative Symptoms Scale | Measured at Baseline and post intervention (6 weeks)
  Measure of negative symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will be shared upon reasonable request

REFERENCES:
- [Background] Granholm E, Holden J, Dwyer K, Mikhael T, Link P, Depp C. Mobile-Assisted Cognitive Behavioral Therapy for Negative Symptoms: Open Single-Arm Trial With Schizophrenia Patients. JMIR Ment Health. 2020 Dec 1;7(12):e24406. doi: 10.2196/24406. PMID 33258792